CLINICAL TRIAL: NCT04757558
Title: C-MAC Video-stylet for Double- Lumen Tracheal Intubation: a Prospective Randomized Study
Brief Title: C-MAC Video-stylet for Double- Lumen Tracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0304793
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Single Lung Ventilation; Thoracic Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC-VS group (Active Comparator): C-MAC-VS will be used to facilitate intubation
  Interventions: Device: C-MAC video-stylet
- control group (Placebo Comparator): direct laryngoscopy using Macintosh laryngoscope will be done for DLT insertion.
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: C-MAC video-stylet — Patients will be randomly assigned two group 40 patients each, C-MAC-VS group (VS group) (Karl Storz GmbHand Co.KG, Germany), and control group (C group). This will be done using a closed envelope technique using a computer-generated block randomization method.
  Arms: C-MAC-VS group
Device: Macintosh laryngoscope — Patients will be randomly assigned two group 40 patients each, C-MAC-VS group (VS group) (Karl Storz GmbHand Co.KG, Germany), and control group (C group). This will be done using a closed envelope technique using a computer-generated block randomization method.
  Arms: control group

SUMMARY:
C-MAC Video Stylet secures the airway. It is a completely new type of video endoscope, it combines the advantages of both rigid and flexible intubation endoscopes. Video allows everyone involved in the intubation to visualize the anatomy simultaneously which facilitates communication and teamwork.

DETAILED DESCRIPTION:
It can be connected easily to the same C- MAC monitor and Pocket Monitor without requiring any additional light source and camera. Video allows everyone involved in the intubation to visualize the anatomy simultaneously which facilitates communication and teamwork. The device has no lumens so it's very easy to clean. Basically if you can get a tube between the cheek and teeth you can intubate the patient.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 years,
* of both sex
* of American Society of Anesthesiologists (ASA) physical Status II and III
* undergoing elective intra-thoracic surgeries requiring double lumen intubation. BMI -< 35 kg/m2,
* with Mallampati score of 1 or 2

Exclusion Criteria:

* Mallampati score > =3;
* inter-incisor distance < 3 cm;
* thyromental distance < 6 cm;
* neck extension < 80°from neck flexion;
* cervical spine instability;
* history of difficult endotracheal intubation
* r difficult mask ventilation; - severe pulmonary ventilation dysfunction
* risk of pulmonary aspiration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
the time taken for intubation (TTI) by C-MAC-VS | 5 minutes
  timing for intubation

CONTACTS AND LOCATIONS:
Overall Officials: rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- rehab Abd Elaziz, Alexandria, Egypt